CLINICAL TRIAL: NCT03951467
Title: Impact of a Strategy Dedicated to Low Health Literacy Level Patients to Improve Their Understanding and Ownership of the Discharge Prescription in Cardio-vascular Diseases
Brief Title: Using an Intervention Adapted to the Health Literacy Level to Improve Adherence to Medical Recommendations
Acronym: ILIADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL19_0035
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Decompensated Heart Failure; Acute Myocardial Infarction
Keywords: Literacy; Cardiovascular Diseases; Interventional study; Randomized Controlled Trial; Tertiary prevention; Health promotion
MeSH Terms: conditions — Literacy; Cardiovascular Diseases | interventions — Health Personnel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental)
  Interventions: Other: Interventional educational toolkit specific to low Health Literacy patients, designed with patients and health professionals.
- Controlled arm (No Intervention): Patients within this arm will be follow as usual care of the cardiologic unit

INTERVENTIONS:
Other: Interventional educational toolkit specific to low Health Literacy patients, designed with patients and health professionals. — Three interviews between the patient and a health advisor trained for the study: two times before discharge from hospital and a telephone reminder within 3 weeks after discharge.
  First and second interview: the nurse will evolve using tools developed in the first phase of the study. The nurse will provide detailed personalized information on the patient's discharge order and illness and the action to be taken depending on the potential situations the patient may encounter.
  Telephone interview: within 3 weeks after discharge, the nurse will repeat the elements of the first interview with the patient to verify that the information has been properly understood and retained and that the patient is able to adopt appropriate behaviors in high-risk situations.
  Two interviews by phone with a clinical reseach assistant at 30 days et 90 days after discharge which consist of questionnaire.
  Arms: Interventional arm

SUMMARY:
Health literacy is the ability to access, understand, evaluate and apply information in order to communicate with health professionals and understand health instructions but also, promote, maintain and improve health throughout life. Health literacy is known as a health determinant. Level of Health Literacy is low or limited within 47% of interrogated people in Europe, resulting in an inability to understand and/or use written texts and digital concepts about one's health.

There is a demonstrated link between low HL and low therapeutic adherence, an increase in the number of re-admissions, and more generally poor health or survival that is even more limited. An association between low LS and higher health care costs has also been reported in the USA and Switzerland. WHO highlight the central role of Health Literacyin health inequalities, regardless of the region of the world.

The investigator chose to conduct this study in patients hospitalized for an acute cardiovascular event: acute myocardial infarction or acute decompensated heart failure , as these patients have cumulative risk factors for misuse and medication errors. They are hospitalized in emergency, for shorter and shorter periods and are discharged with complex drug treatments. The data show that the return home after acute hospitalization for these conditions is a particularly high-risk period for medication errors and misuse, especially with low level of Health Literacy. The proportion of patients with preventable adverse events in the weeks following their return home ranges from 23% to 30% and nearly 60% are re-hospitalized within 6 months.

The hypothesis of the study is that in patients hospitalized for cute myocardial infarctionor acute decompensated heart failurewith low Health Literacy levels, information on discharge treatment using appropriate tools and techniques will reduce the risk of patient-related medication errors or misuse within 30 days of discharge.

The purpose of this study is to develop an educational intervention model adapted to low Health Literacy levels and routinely feasible, even in case of short stays, in complementarity with traditional therapeutic education programmes that require higher investments and are therefore not accessible to all patients. This innovative approach could then be applied to a large number of chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Hospitalization for at least a 2nd acute attack (systolic or diastolic)
* Patient living at home before hospitalization for decompensation
* Affiliated with a health insurance plan

Exclusion Criteria:

* Short-term vital prognosis
* Bipolar disorders, active psychoses
* Severe dementia
* Psychiatric or cognitive comorbidities making inclusion impossible, at the discretion of the investigator.
* Pregnant, parturient or breastfeeding women
* Persons deprived of liberty by a judicial or administrative decision
* Persons admitted to a health or social establishment for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Subject participating in another interventional research including an exclusion period still ongoing at inclusion
* Score S-TOFHLA (>22)
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-12-26 (Estimated); Study Completion 2027-12-26 (Estimated)

PRIMARY OUTCOMES:
Patient-related medication errors or misuse within 30 days of discharge from hospital. | Day 30
  This criterion is defined as the proportion of patients who have made a medication error or misuse, with or without a clinical consequence.
  We will focus on patient-related medication errors and misuse, i.e. non-compliance with prescription (shorter or longer treatment time, dosage changes, self-medication, etc.), based on the definition proposed by Kripalani et al.
  An adjudication committee composed of three independent experts will be responsible for defining the potential severity of drug errors or misuses related to the main judgement criterion.
  Data on primary endpoint will be collected by a clinical researcher, blinded to the randomization group, using a standardized questionnaire administered during the 30-day telephone interview. The patient will be asked the names of the treatments, how he/she took them (number of units per intake, frequency of intake,...), self-medication taken and medical follow-up (medical consultations, biological follow-up,...) over the past 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Julie HAESEBAERT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (4):
- France (4):
  - Hôpital Louis Pradel, Bron
  - Public Health Department, Lyon
  - Hôpital Lyon Sud, Pierre-Bénite
  - SSR Val Rosay, Saint-Didier-au-Mont-d'Or

IPD SHARING:
Plan to Share IPD: No